CLINICAL TRIAL: NCT01619449
Title: Continuous Renal Replacement Therapy in the Setting of Orthotopic Liver Transplant: A Randomized Trial
Brief Title: Continuous Renal Replacement Therapy in the Setting of Orthotopic Liver Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research never begun and no subjects enrolled. Protocol term with IRB in Dec 2014
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #11-0626
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Acute Kidney Injury; Liver Disease; Chronic Kidney Disease; End Stage Kidney Disease
Keywords: Acute Kidney Injury; Continuous Renal Replacement Therapy; Liver Transplant
MeSH Terms: conditions — Acute Kidney Injury; Liver Diseases; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal replacement therapy (Experimental): Liver transplant recipients who receive continuous renal replacement therapy intra-operatively.
  Interventions: Procedure: Renal replacement therapy
- No CRRT (Active Comparator): This arm consists of standard of care without CRRT in the OR for OLT
  Interventions: Procedure: Renal replacement therapy

INTERVENTIONS:
Procedure: Renal replacement therapy — Liver transplant recipients receiving continuous renal replacement therapy for duration of liver transplant surgery.

SUMMARY:
To evaluate the efficacy of continuous renal replacement therapy (CRRT) during orthotopic liver transplantation (OLT) in clearing excess solutes and improving acid-base parameters. The investigators hypothesize that the use of intra-operative CRRT in OLT recipients is associated with increased solute removal and improved acid-base statues when compared to controls who do not receive CRRT

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and able to sign consent (or surrogate)
* Receiving liver or combined liver-kidney transplant
* eGFR < or equal to 40 ml/min immediately prior to transplant or currently on any form of renal replacement therapy for acute kidney injury or end-stage renal disease
* Pre-operative potassium of < or equal to 5.5 mEq/L

Exclusion Criteria:

* Pre-operative hemoglobin < or equal to 7 g/dL
* Pre-operative weight > or equal to 125 kig

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Solute Clearance | Intra-operative time
  To compare the clearance of solutes (ie. potassium, lactate, creatinine and blood urea nitrogen) by CRRT in renally impaired OLT recipients to OLT recipients who do not receive CRRT

SECONDARY OUTCOMES:
Renal function and patient outcomes | 1 year post-operatively
  To compare long-term maintenance of renal function (12 months) and other health outcomes in OLT recipients who received CRRT versus OLT recipients who did not receive OLT

CONTACTS AND LOCATIONS:
Overall Officials: Jay L Koyner, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States